CLINICAL TRIAL: NCT07201142
Title: Gingival Crevicular Fluid and Salivary Levels of GDF-15, Smad2, Smad5, Smad6, and IL-6 in Patients With Periodontitis
Status: Completed | Type: Observational
Sponsor: Melis Yilmaz (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor-Investigator, Melis Yilmaz, Dr., Medipol University
Organization: Medipol University (Other)
Other Study IDs: 1097/22.12.2022
Record Dates: First submitted 2025-05-30; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis; Periodontal Disease
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis
- Control: Periodontally Healthy

SUMMARY:
The dysregulation of the transforming growth factor-beta signaling pathway can lead to inflammation and tissue destruction in the pathogenesis of periodontitis. This study aims to evaluate the levels of GDF-15, Smad 2, Smad 5, Smad 6, and IL-6 in gingival crevicular fluid (GCF) and saliva between individuals with periodontitis and periodontal healthy controls and to evaluate the relationship of these biomarkers with clinical periodontal parameters. This study aims to investigate the levels of GDF-15, Smad2, Smad5, Smad6, and IL-6 in GCF and saliva samples from individuals with periodontitis and periodontally healthy controls, as well as to assess the associations of these biomarkers with clinical periodontal parameters. A total of 44 systemically healthy individuals, including 22 patients diagnosed with stage III/grade B periodontitis and 22 periodontal healthy individuals, were included in the study. Clinical periodontal parameters (plaque index (PI), probing depth (PD), clinical attachment level (CAL), and bleeding on probing (BOP)) were recorded. GDF-15, Smad 2, Smad 5, Smad 6, and IL-6 levels in saliva and GCF were analyzed using the ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years of age;
* having at least 20 natural teeth excluding third molars;
* being systemically healthy

Exclusion Criteria:

* under 18 years of age;
* had used antibiotics
* had used nonsteroidal anti-inflammatory drugs, corticosteroids, immunosuppressants, beta-blockers, calcium channel blockers, anticoagulants, or hormonal contraceptives within the past 6 months;
* had systemic diseases such as diabetes mellitus, rheumatoid arthritis, cardiovascular diseases, epilepsy, renal or hepatic disorders, or viral infections like HIV/AIDS;
* pregnant or breastfeeding;
* current smokers or had a history of alcoholism;
* had received nonsurgical periodontal therapy within the last 6 months or surgical periodontal treatment within the last 12 months;
* had fewer than 20 natural teeth (excluding third molars);
* had fixed orthodontic appliances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprised individuals who presented to the Department of Periodontology at Istanbul Medipol University between April and October 2023 for dental consultation or treatment.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
GCF GDF-15, GCF IL-6, GCF SMAD 2, GCF Smad 5, GCF Smad 6 | September 2023 to February 2024
Saliva GDF-15, Saliva IL-6, Saliva SMAD 2, Saliva Smad 5, Saliva Smad 6, | September 2023 to Februart-y 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No